CLINICAL TRIAL: NCT06965374
Title: Foslevodopa/Foscarbidopa REal-world Evidence in Parkinson's Disease Quality of LIFE Outcomes
Brief Title: Real-World Study of Foslevodopa/Foscarbidopa to Assess Quality of Life Outcomes in Adult Participants With Advanced Parkinson Disease
Acronym: FREELIFE
Status: Recruiting | Type: Observational
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Other Study IDs: P25-246
Record Dates: First submitted 2025-05-02; First posted 2025-05-11 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Parkinson Disease
Keywords: Parkinson Disease; Foslevodopa/Foscarbidopa
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Foslevodopa/Foscarbidopa: Participants will receive Foslevodopa/Foscarbidopa as prescribed by their physician according to local label.

SUMMARY:
Parkinson's disease (PD) is a neurological condition, which affects the brain. PD gets worse over time, but how quickly it progresses varies a lot from person to person. Some symptoms of PD are tremors, stiffness, and slowness of movement. This study will assess how effective Foslevodopa/Foscarbidopa is in treating Italian adult participants with advanced Parkinson disease under routine clinical practice. This study will also assess the caregiver quality of life (QOL) (if caregiver is present).

Foslevodopa/Foscarbidopa is an approved drug for the treatment of Parkinson's Disease. Approximately 270 adult participants who are prescribed Foslevodopa/Foscarbidopa by their doctors will be enrolled across approximately 19 sites in Italy.

Participants will receive Foslevodopa/Foscarbidopa subcutaneous infusion as prescribed by their physician. Participants will be followed for up to 12 months.

There is expected to be no additional burden for participants in this trial. Participants will attend regular visits during the study at a hospital or clinic according to their routine clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Participants with a diagnosis of levodopa-responsive advance Parkinson's disease (PD)
* Investigator decision on participant treatment with subcutaneous Foslevodopa/Foscarbidopa (LDp/CDp) made prior to, and independently, the decision to approach the participant to participate in the study
* 24-h subcutaneous LDp/CDp treatment prescribed in accordance with the applicable approved label and local regulatory and reimbursement policies

Exclusion Criteria:

* Any condition included in the contraindications section of the approved local subcutaneous LDp/CDp label
* Participation in a clinical trial of an investigational drug, concurrently or within the last 30 days. Participation in another Post-Marketing Observational Study (PMOS) or Registry is acceptable
* History of relevant skin conditions or disorders (e.g., psoriasis, atopic dermatitis) per investigator´s judgment. In case of temporary affections like recent sunburn, acne, scar tissue, tattoo, open wound, branding, or colorations, the subject should not be included if the investigator considers these as interfering with the infusion of study drug or with study assessments

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with advanced Parkinson disease treated with Foslevodopa/Foscarbidopa according to label in Italy
Sampling Method: Non-Probability Sample
Enrollment: 270 (Estimated)
Dates: Start 2025-06-04 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Change From Baseline in Quality of Life as Measured by PD Questionnaire-39 (PDQ-39) Summary Index | Up to approximately 6 months
  The PDQ-39 is a self-administered questionnaire which comprises 39 items addressing 8 domains of health in PD. These include: mobility, activities of daily living, emotional well-being, stigma, social support, cognition, communication, and bodily discomfort. The total score is between 0 and 156, calculated as the total sum of the items, and higher scores are associated with more severe symptoms. Negative changes from baseline indicate improvement.

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (17):
- Italy (17):
  - IRCCS Oasi SS. Troina /ID# 273507, Troina, Enna
  - Istituto Neurologico Mediterraneo Neuromed S.P.A. - Irccs /Id# 272695, Pozzilli, Isernia
  - ASST Centro Specialistico Ortopedico Traumatologico Gaetano Pini-CTO /ID# 272949, Milan, Milano
  - Fondazione IRCCS Istituto Neurologico Carlo Besta /ID# 273225, Milan, Milano
  - Azienda Ospedaliera Universitaria Luigi Vanvitelli /ID# 273434, Naples, Napoli
  - A.O.U. CITTA' DELLA SALUTE E DELLA SCIENZA DI TORINO - Ospedale Molinette /ID# 273276, Turin, Piedmont
  - Azienda Ospedaliera Universitaria Policlinico Tor Vergata /ID# 272834, Rome, Roma
  - Azienda Ospedaliero-Universitaria Policlinico Umberto I /ID# 273562, Rome, Roma
  - Fondazione Policlinico Universitario Agostino Gemelli IRCCS-Universita Cattolica /ID# 274539, Rome, Roma
  - Azienda Ulss 3 Serenissima /ID# 273027, Venice, Venezia
  - Azienda Ospedaliero Universitaria delle Marche /ID# 272694, Ancona
  - IRCCS Centro Neurolesi Bonino Pulejo /ID# 273628, Messina
  - Azienda Ospedale-Universita Padova /ID# 274317, Padua
  - Azienda Ospedaliera Universitaria Policlinico Paolo Giaccone /ID# 272863, Palermo
  - Fondazione Mondino Istituto Neurologico Nazionale a Carattere Scientifico IRCCS /ID# 274226, Pavia
  - AUSL di Reggio Emilia - Arcispedale Santa Maria Nuova /ID# 274388, Reggio Emilia
  - AOU San Giovanni di Dio Ruggi d'Aragona - Scuola Medica Salernitana /ID# 274319, Salerno

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Related Info — https://www.abbvieclinicaltrials.com/study/?id=P25-246